CLINICAL TRIAL: NCT05866692
Title: A Phase I, Multicenter, Open-label Study of TY-2699a, Administered Orally in Adult Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of TY-2699a in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: TYK Medicines, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TYKM1805102
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TY-2699a (Experimental): Escalation stage: Multiple doses of TY-2699a as monotherapy for oral administration to find the maximum tolerated dose.
  Expansion stage: an optimal dose of TY-2699a for cohort expansion.
  Interventions: Drug: TY-2699a

INTERVENTIONS:
Drug: TY-2699a — TY-2699a PO, BID
  Escalation stage: increased dose cohorts from low dose to MTD
  Expansion stage: The dose for the Expansion stage will be determined based on results

SUMMARY:
This is a phase I, multicenter, open-label study. The study will investigate the safety, tolerability, PK, and preliminary efficacy of TY-2699a on locally advanced or metastatic solid tumors.

DETAILED DESCRIPTION:
To assess the safety and tolerability of TY-2699a when administered as a single agent in subjects with locally advanced or metastatic solid tumors.

To determine the maximum tolerated dose (MTD), and the recommended phase 2 dose (RP2D) as a single agent in subjects with locally advanced or metastatic solid tumors.

To evaluate the pharmacokinetics (PK) of TY-2699a administered at single and multiple oral doses.

To assess the preliminary antitumor activity of TY-2699a as a single agent in subjects with locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to provide written informed consent approved by institutional review board (IRB) or independent ethics committee (IEC).
2. Age ≥18 years.
3. At the escalation stage, patients should fulfill the following criteria at Screening:

1) Participants with locally advanced or metastatic solid tumors including TNBC, ER+HER2-BC, ovarian cancer, small cell lung cancer, castrate-resistant prostate cancer (CRPC), or PDAC with KRAS mutant; Or any other locally advanced or metastatic solid tumor with evidence of deregulated RB-pathway based on available molecular test results and after sponsor review to confirm eligibility as determined with prior molecular assays performed in a CLIA-certified or equivalent laboratory. (Note: ① 0% - 1% of tumor cells expressing ER or PR as negative while ≥ 1% of tumor cells expressing ER or PR as positive on IHC staining, recommended by ASCO/CAP guideline Update 2020; negative HER2 is defined as IHC 0 or 1+, or IHC 2+ but confirmed by the negative ISH, recommended by ASCO/CAP Guideline 2018; ② Genes of KRAS and other biomarkers will be detected by the Polymerase Chain Reaction (PCR) or Next-Generation Sequencing (NGS)); 2) Patients who have progressed on established standard medical anti-cancer therapies for a given tumor type or have been intolerant to such therapy, or in the opinion of the investigator have been considered ineligible for a particular form of standard therapy on medical grounds.

4. At the expansion stage, patients should fulfill the following criteria at Screening :

1)Cohort : TNBC patients progressed on ≥ 2 previous lines of therapy and/or other solid tumors will receive TY-2699a. ① Previous therapy can be of any nature (chemotherapy, immunotherapy, antiangiogenics, experimental therapy, etc.); ② Histologically-confirmed breast carcinoma not expressing ER, PR, and HER2 (negative ER and PR is defined as < 1% tumor cells expressing ER and PR on IHC staining, recommended by ASCO/CAP Guideline Update 2020; negative HER2 is defined as IHC staining 0 or 1+ , or IHC 2+ but confirmed by the negative ISH, recommended by ASCO/CAP Guideline 2018; negative HER2 is defined as IHC 0 or 1+, or IHC 2+ but confirmed by the negative ISH, recommended by ASCO/CAP Guideline 2018); ③ With or without BRCA mutation.

5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1, and life expectancy > 3 months.

6. Capability to swallow intact capsule (without chewing, crushing or opening). 7. At least 1 measurable target lesion according to Response Evaluation Criteria in Solid Tumor Version 1.1 (RECIST v1.1, Appendices 15.2 RECIST v1.1 ) determined by the investigator.

8. All acute toxic effects (excluding alopecia and neuropathy associated with prior platinum-based drug therapy) of any prior therapy recovered to grade ≤1 based on NCI CTCAE v5.0.

9. Baseline laboratory results fulfilling the following requirements: Absolute neutrophils count (ANC) ≥1500/mm3 (1.5×109/L) * Platelets ≥100,000/mm3 (100×109/L) * Hemoglobin > 90 g/L* Estimated creatinine clearance ≥55 mL/min+ Total serum bilirubin <1.5 × ULN <3.0 × ULN if known Gilbert's disease Liver transaminases (AST/ALT) <2.5 × ULN; <5 × ULN if liver metastases are present ULN: upper limit normal.

* No blood transfusion, blood products, or hematopoietic factors such as G-CSF, erythropoietin or albumin within 14 days prior to first dose.

  * Cockcroft-Gault Equation. 10. For female patients of childbearing potential, the serum or urine pregnancy test within 7 days prior to the start of TY-2699a treatment should be negative.

    11. Male and female patients of childbearing potential must agree to use at least two method of highly effective contraception from signing ICF, throughout the study and continued for 90 days after the last dose of TY-2699a treatment at the escalation stage or for the labeled duration of contraception of the combined approved drug fulvestrant (e.g., FASLODEX requires one-year contraception after the last dose) or PD-L1 antibody (will decide a brand approved in US before starting expansion stage) after the last dose at the expansion stage.

    12. Willing and able to comply with all aspects of the protocol.

Exclusion Criteria:

1. Concurrent participation in another interventional clinical trial, unless the patient at long-term follow-up period.
2. Patients with the following treatment:

   1. Received undergone major surgery (except minor surgery such as appendicitis, tumor biopsy, etc.) within 4 weeks prior to the first dose.
   2. Received bone marrow (equal to area of pelvis) or extensive radiation therapy within 28 days prior to the first dose; received local radiation therapy (e.g., thoracic spine and rib radiation therapy) within 7 days prior to the first dose of the study drug.
   3. Received CYP3A and CYP2C8 strong inducers/strong inhibitors or p-gp glycoprotein inhibitors within 14 days prior to the first dose (see Appendices 15.3 Examples of CYP450-related Drugs/food).
   4. History of proton pump inhibitors (PPIs) within 4 days prior to the first dose of TY-2699a; OR history of histamine H2 blockers within 2 days prior to the first dose of TY-2699a. Patients who are receiving and require continuation of drug therapy during the study with drugs known to prolong the QTc interval or that may cause torsades de pointes.
   5. Prior exposure to transcriptional kinase family CDK inhibitors, such as the CDK7 and CDK9 inhibitors SY-5609，CT-7001，Alvocidib，Dinaciclib，Seliciclib and SY-1365. Exception: Previous exposure to cell cycle CDK inhibitors such as inhibitors of CDK4 and CDK6 (ie, palbociclib) is allowed.
3. History of other previous cancer (except for squamous cell or basal-cell carcinoma of the skin, or any in situ carcinoma that has been completely resected), requiring therapy within the previous 5 years
4. Patients with unstable brain metastases: Patients with CNS complications requiring urgent neurosurgical treatment (e.g., surgery, etc.) (except when surgery is completed >7 days and side effects from complications are ≤ grade 1); patients requiring glucocorticoids, mannitol or diuretics at equivalent doses greater than 4 mg of dexamethasone to control symptoms of brain metastases within 14 days prior to the first study dose; patients who have undergone whole brain radiation therapy or gamma knife within 14 days prior to the first study dose; patients with symptoms of spinal cord compression from the tumor. Note: conversely, patients with stable CNS metastasis and those who are beyond the treatment washout period of 14 days per protocol are eligible to the study.
5. Epilepsy needing treatment; having a history of psychotropic substance abuse that cannot abstain; have mental disorders (successful abstain must pass at least 2 weeks without observing withdrawal reaction).
6. Patients receiving long-term systemic immunosuppressant therapy (≤10 mg/ day of prednisone or other equivalent dose of corticosteroid inhalation or topical administration can be included).
7. Any of the following cardiac criteria:

   1. Mean resting corrected QT interval (electrocardiogram interval measured from the onset of the QRS complex to the end of the T wave) for heart rate QTc > 470 msec obtained from 3 electrocardiograms, using the screening clinic electrocardiogram machine derived QTc value.
   2. Any clinically important abnormalities in rhythm, conduction, or morphology of resting electrocardiogram (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval >250 msec). Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or any concomitant medication known to prolong the QT interval during Screening.
   3. Left ventricular ejection fraction (LVEF) <50%；
   4. Clinically significant cardiovascular disease (either active at Screening or within 6 months prior to enrollment): myocardial infarction, unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure (New York Heart Association Classification Class ≥II), cerebrovascular accident or transient ischemic attack, stroke, symptomatic bradycardia, or requirement for anti-arrhythmic medication.
   5. Unstable patients that may affect their safety or compliance of study, any serious or uncontrolled systemic disease including uncontrolled high blood pressure (systolic blood pressure >160mmHg, or diastolic pressure >100mmHg), uncontrolled diabetes (fasting plasma glucose >10 mmol/L), active bleeding, severe eye disease, severe psychosis, nerve, vascular, or respiratory disease.
8. Known active infections, including human immunodeficiency virus (HIV), hepatitis B virus (HBV), and hepatitis C virus (HCV) infection, except for asymptomatic chronic HBV or HCV carriers. Active HBV, HCV, or HIV infections are defined as

   1. Hepatitis B surface antigen (HBsAg) positive and HBV-DNA ≥ 2000 cps/mL or 500 IU/mL; HBsAg-negative, anti-HBc-positive patients are at high risk of HBV reactivation who require suppressive antiviral therapy prior to initiation of cancer therapy
   2. Anti-HCV antibody positive and HCV-RNA > upper normal limit defined by sites
   3. Anti-HIV antibody positive with uncontrolled opportunistic infections; anti-HIV antibody positive with CD4+ count < 350 cells/uL that requires HIV therapy prior to the cancer treatment; other conditions allowing concurrent ART but the therapy not tolerated and that the toxicities confused with investigational drug toxicities. Note: Examples of drug-drug interactions that affect absorption, distribution, metabolism, and excretion of the TY-2699a are shown in Appendices 15.3 Examples of CYP450-related Drugs/food.
9. Diagnosed interstitial lung disease with or without symptoms, as well as conditions that may cause pulmonary toxicity or related pneumonia after using TY-2699a, or pulmonary symptoms deemed by the investigator to have high risk of developing interstitial lung disease. Note: Patients with history of prior radiation pneumonitis will not be excluded.
10. Active gastrointestinal disease with significant symptoms (e.g., gastric ulcer, Crohn's disease, ulcerative colitis, short gut syndrome) or other malabsorption syndromes that will impact in ingesting, transporting, or absorbing the drug.
11. Known/suspected allergy to the composition of TY-2699a or the analogues.
12. Pregnant and breastfeeding women.
13. The Prinicpal Investigator considers that the patient is not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Escalation stage) Dose Limiting Toxicities (DLTs) | Within 28 days of the first dose
  Numbers of participants experiencing AEs which are defined as DLTs classfied by CTCAE v5.0.
(Escalation stage) Recommended Phase 2 Dose (RP2D) | Within 28 days of the last patient dosed in escalation stage
  The RP2D is defined as the dose level chosen for the dose expansion arms, based on safety, tolerability, efficacy, pharmacokinetics (PK), and pharmacodynamic (PD) data collected during the dose escalation portion of the study.
(Escalation stage) Adverse events (AEs) | From Baseline up to 28 days after the end of the treatment
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.
(Expansion stage) Overall Response Rate (ORR) | From the date of first dose until the date of first documented progression or stable disease or the date of death from any cause, whichever came first, assessed up to 30 months.
  ORR is defined as the percentage of subjects who have a partial response (PR) or complete response (CR) to the treatment response assessment in accordance to Response Evaluation Criteria in Solid Tumors (RECIST 1.1).

SECONDARY OUTCOMES:
(Escalation and Expansion stage) Area under the plasma concentration time curve(AUC0-inf) | Cycle 1 Day 1 (at pre-dose) and Cycle 1 Day 28 (at pre-dose, 0.5, 1, 2, 4, 8, 12 hours post-dose)(Each Cycle=28 days)
  AUC0-inf defined as the area under the plasma concentration-time curve from time 0 extrapolated to Infinite time.
(Escalation and Expansion stage) Area under the plasma concentration time curve(AUC0-t) | Cycle 1 Day 1 (at pre-dose) and Cycle 1 Day 28 (at pre-dose, 0.5, 1, 2, 4, 8, 12 hours post-dose)(Each Cycle=28 days)
  AUC0-t defined as area under the plasma concentration-time curve from time 0 to time t.
(Escalation and Expansion stage) Maximum plasma concentration (Cmax) | Cycle 1 Day 1 (at pre-dose) and Cycle 1 Day 28 (at pre-dose, 0.5, 1, 2, 4, 8, 12 hours post-dose)(Each Cycle=28 days)
  Cmax is the maximum (or peak) plasma concentration that the drug achieves in blood after the drug has been administered.
(Escalation and Expansion stage) Minimum plasma concentration (Cmin) | Cycle 1 Day 1 (at pre-dose) and Cycle 1 Day 28 (at pre-dose, 0.5, 1, 2, 4, 8, 12 hours post-dose)(Each Cycle=28 days)
  Cmin is the minimum plasma concentration that the drug achieves in blood after the drug has been administered.
(Escalation and Expansion stage) The time to the peak concentration (Tmax) | Cycle 1 Day 1 (at pre-dose) and Cycle 1 Day 28 (at pre-dose, 0.5, 1, 2, 4, 8, 12 hours post-dose)(Each Cycle=28 days)
  Tmax is defined as the time of maximum concentration of the drug in blood observed after a drug dose administration.
(Escalation and Expansion stage) Progression-free survival (PFS) | Up to 30 months after the date of first dose.
  PFS is defined as the time from randomization until first evidence of disease progression or death.
(Escalation and Expansion stage) Duration of Response (DOR) | Up to 30 months after the date of first dose.
  DOR is defined as the time from randomization to disease progression or death in patients who achieve complete or partial response.
(Escalation and Expansion stage) Overall survival (OS) | Up to 30 months after the date of first dose.
  OS is defined as the time from the start of treatment to death or the end of the study.
(Escalation stage) Overall Response Rate (ORR) | From the date of first dose until the date of first documented progression or stable disease or the date of death from any cause, whichever came first, assessed up to 30 months.
  ORR is defined as the percentage of subjects who have a partial response (PR) or complete response (CR) to the treatment response assessment in accordance to Response Evaluation Criteria in Solid Tumors (RECIST 1.1).

CONTACTS AND LOCATIONS:
Overall Officials: TYK Medicines, Inc, Study Director — TYK Medicines, Inc
Locations (2):
- China (2):
  - National Cancer Center/Cancer Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Beijing, Beijing Municipality
  - Shandong Cancer Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No